CLINICAL TRIAL: NCT00803257
Title: Effect of Lumbrical Stretching on Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Nancy Baker, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 07030166
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Splint; Hand exercises
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Lumbrical splint and lumbrical stretches
  Interventions: Other: Lumbrical splint and Lumbrical exercises
- 2 (Active Comparator): Lumbrical Splint and regular exercises
  Interventions: Other: Lumbrical splint and Lumbrical exercises
- 3 (Active Comparator): Regular splint and lumbrical exercises
  Interventions: Other: Lumbrical splint and Lumbrical exercises
- 4 (Active Comparator): Regular splint and regular exercises
  Interventions: Other: Lumbrical splint and Lumbrical exercises

INTERVENTIONS:
Other: Lumbrical splint and Lumbrical exercises — Subjects receive one of four possible interventions - Dose and Frequency are the same for each

SUMMARY:
Symptoms of CTS occur when any condition decreases the size of the carpal canal or increases the volume of the structures within the carpal canal, compressing the median nerve. One cause of the symptoms of CTS is the incursion of the lumbrical muscles of the hand into the carpal canal. Individuals with CTS tend to have tight lumbrical muscles which increase this incursion, thereby increasing CTS symptoms. An intervention designed to reduce the incursion of the lumbrical muscles should have an effect on the symptoms of CTS.

The purpose of this study is to systematically examine the effect of an intensive lumbrical muscle intervention, splinting to prevent lumbrical muscle incursion and lumbrical muscle exercises, on the symptoms of CTS. This project will be a randomized clinical trial to evaluate the effectiveness of a home program targeting the lumbrical muscles. One hundred and twenty subjects will be assigned to one of 4 groups: Group 1 will receive a home program of lumbrical muscle stretches combined with a lumbrical positioning splint; Group 2 will receive a home program of lumbrical muscle stretches combined with a night wrist cock-up splint; Group 3 will receive a home program of general stretches combined with a lumbrical positioning splint; and Group 4 will receive a home program of general stretches combined with a night wrist cock-up splint. After 1 month, 3 months, and 6 months the groups will be compared to determine if there is a significant reduction in symptoms between the groups.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 yo
* Clinical symptoms of Carpal tunnel syndrome (CTS)
* Positive Tinel's, Phalen's, or Durkin's test
* Absence of thenar atrophy
* 2 pt discrimination of 5mm or less

Exclusion Criteria:

* Persons needing immediate CTS surgery
* Pregnancy
* Compressive neuropathy in the ipsilateral arm
* Diabetes
* prior CTS release
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Carpal Tunnel Syndrome Symptom Severity and Functional Status Scale (CTS-SSFS) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Baker NA, Moehling KK, Desai AR, Gustafson NP. Effect of carpal tunnel syndrome on grip and pinch strength compared with sex- and age-matched normative data. Arthritis Care Res (Hoboken). 2013 Dec;65(12):2041-5. doi: 10.1002/acr.22089. PMID 23925936
- [Derived] Baker NA, Moehling KK, Rubinstein EN, Wollstein R, Gustafson NP, Baratz M. The comparative effectiveness of combined lumbrical muscle splints and stretches on symptoms and function in carpal tunnel syndrome. Arch Phys Med Rehabil. 2012 Jan;93(1):1-10. doi: 10.1016/j.apmr.2011.08.013. PMID 22200381